CLINICAL TRIAL: NCT04093310
Title: Cost-utility Analysis Treatment of Bartholin's Abscess : Word Catheter Versus Incision-drainage.
Acronym: BARTHO-KT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC19_0179
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Bartholin's Gland Abscess Treatment
Keywords: incision-drainage; Bartholin's abscess; Word catheter; Marsupialization; Cost-utility analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Word catheter (Experimental): The abscess is incised and the Word catheter is inserted into the residual cavity to create a neo-channel to prevent recurrence. The catheter is removed after 4 weeks during a consultation
  Interventions: Device: Word Catheter
- Incision-drainage (Active Comparator): This procedure performed under general or loco-regional anaesthesia consists in incising the abscess, draining the pus build-up and placing a wick in the residual cavity to promote progressive healing from the inside out.
  Interventions: Procedure: Incision-drainage

INTERVENTIONS:
Device: Word Catheter — Use of the Word catheter to remove the Bartholin's abscess
  Arms: Word catheter
Procedure: Incision-drainage — Incision-drainage to remove the Bartholin's abscess
  Arms: Incision-drainage

SUMMARY:
Bartholin's gland abscess is a condition requiring emergency consultation. Placement of a Word catheter, which is a minor technique used in France as a treatment of bartholin's Abscess, can be done in an emergency room without hospitalization. Actually, incision-drainage, which is the most widespread treatment in France, is performed on day surgery with or without overnight hospitalization. Our hypothesis is that the use of Word catheter compared to incision-drainage would not modify the quality of life of the patients but would allow a saving of up to 3 M€ per year in France.

ELIGIBILITY:
Inclusion Criteria:

Abscess of Bartholin's gland Patient able to understand the protocol Patient who signed informed consent Patient with social insurance

Exclusion Criteria:

Spontaneous fistulization of the abscess before surgical treatment Abscess volume under 3 ml Medical treatment which avoid incision or word catheter placement patients under guardianship Unable to complete questionnaires Patients not affiliated to social protection regimen Pregnant or post-partum women (until 4 weeks after delivery)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
cost-utility ratio, according to the societal perspective of the of the management of Bartholin's gland abscess by the Word catheter compared to the incision-drainage | 12 months
  The utility will be measured by:
  Quality Adjusted Life Year (QALYs) as estimated from responses to the Euroqol-5 Dimensions (EQ-5D 5L) health-related quality of life questionnaire. The questionnaire focuses on 5 dimensions: mobility, personal autonomy, current activities, pain/discomfort and anxiety/depression. For each of these dimensions, 5 answers are possible.
  The costs will be measured by the addition of the following costs:
  Outpatient resource consumption collected in a declarative patient questionnaire. Hospital care resources using the the database of the Medicalised Information System Program of each recruiting site

SECONDARY OUTCOMES:
Budget impact analysis for the health insurance point of view in case of diffusion of the Word catheter | 5 years
  Comparison of intervention costs on the study sample and projection of these costs over 5 years, from the health insurance and hospital perspectives
Non inferiority evaluation of Word catheter vs. Incision drainage in terms of pain | at baseline and day 1
  Pain numeric scale from 0 to 10
Non inferiority evaluation of Word catheter versus incision-drainage in terms of recurrence rate | 12 months
  Number of homolateral recurrences of Bartholin's abscess, declared by the patient
Comparison of Word catheter versus incision-drainage concerning pain | 12 months
  Pain numeric scale from 0 to 10
Comparison of Word catheter versus incision-drainage concerning management time | Day 0 (procedure day), Day 1
  Date and time of patient initial management (randomization) Date and time of the beginning of the procedure date and time of the end of the procedure date and time of the hospital departure
Comparison of Word catheter versus incision-drainage in terms of complications | 12 months
  number of complications related to the procedure (healing complications, infection, lost of the Word catheter), contro-lateral Bartholin's abscess occurrence
Comparison of Word catheter versus incision-drainage in terms of surgical failure | Immediate post-operative (D0) and one month
  Word catheter: insertion failure, loss, removal decision (from the patient or the surgeon) Incision-drainage: incomplete drainage
Comparison of Word catheter versus incision-drainage in terms of impact on sexual activity | Baseline, one month, 6 months and 12 months
  Score of the Female Sexual Function Index: self-questionnaire including 19 questions assessing different parameters of the sexual activity
Comparison of Word catheter versus incision-drainage in terms of quality of life using the SF-12-HS | Baseline, one month, 6 months and 12 months
  Short-Form-12-Health-Survey questionnaire score: self-questionnaire including 12 questions measuring different aspects of quality of life
Comparison of Word catheter versus incision-drainage in terms of quality of life using the EQ-5D | Baseline, one day, one month, 3 months, 6 months, 9 months and 12 months
  EQ-5D 5L score (described in primary outcome)
Comparison of Word catheter versus incision-drainage in terms global patient impression and improvement | One day, one month, 3 months, 6 months, 9 months and 12 months
  Patient Global Impression and Improvement (PGI-I) global index used to rate the response of a condition to a therapy (transition scale). It is a single question asking the patient to rate their global condition now, as compared with how it was prior to before beginning treatment on a scale from 1 - very much better to 7 - very much worse

CONTACTS AND LOCATIONS:
Overall Officials: Thibault Thubert, PhD, Principal Investigator — Nantes University Hospital
Locations (17):
- France (17):
  - Chu Angers, Angers
  - Bordeaux University Hospital, Bordeaux
  - CHU CAEN, Caen
  - Ch Antoine Beclere, Clamart
  - Chu Estaing, Clermont-Ferrand
  - Institut Franco Britannique, Levallois-Perret
  - Chu Lille, Lille
  - Nancy University Hospital, Nancy
  - Chu Nantes, Nantes
  - Chu Caremeau, Nîmes
  - Ch Kremlin Bicetre, Paris
  - Chu Cochin, Paris
  - Chu Robert Debre, Paris
  - Chi Poissy, Poissy
  - Chu Poitiers, Poitiers
  - Rennes University Hospital, Rennes
  - Chu Toulouse, Toulouse